CLINICAL TRIAL: NCT06940427
Title: Development of FAPI PET as a Non-invasive Biomarker of Pulmonary Fibrogenesis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-0489; A539300 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison); Protocol Version 3/27/25 (Other: UW Madison)
Record Dates: First submitted 2025-04-14; First posted 2025-04-23 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Fibrosis Lung
Keywords: lung disease associated with fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Groups A and B will be parallel; however, Group B participants will have the option to crossover to Group A upon completing Group B participation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Group A - 3 scans (Experimental): Participants undergo three PET/MRI scans using the FAPI radiotracer. They will have 3 research visits, and each visit may last up to 2.5 hours.
  Interventions: Drug: FAPI tracer; Device: PET/MRI
- Group B - 2 scans (Experimental): Participants undergo two PET/MRI scans using the FAPI radiotracer. They will have 2 research visits, and each visit may last up to 2.5 hours.
  Interventions: Drug: FAPI tracer; Device: PET/MRI
- Group B Crossover (Experimental): Participants undergo two additional PET/MRI scans using the FAPI radiotracer. They will have 2 additional research visits, and each visit may last up to 2.5 hours.
  Interventions: Drug: FAPI tracer; Device: PET/MRI

INTERVENTIONS:
Drug: FAPI tracer — radioactive substance called a "tracer" injected into the arm
Device: PET/MRI — positron emission tomography (PET) takes pictures of inside of the body

SUMMARY:
The goal of this clinical trial is to gain more information about how fibroblast activation protein inhibitor (FAPI) binds to a certain type of cells in fibrotic lung tissue and how this information can be used to better diagnose and track fibrotic lung disease activity.

Participants will undergo up to 4 PET/MRI scans using the FAPI radiotracer.

DETAILED DESCRIPTION:
Researchers aim to develop a non-invasive PET/MRI imaging tool using FAPI as a PET radiotracer and MRI to assess the presence and extent of fibrogenesis (the process that leads to fibrosis and scarring) in the lungs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able and willing to provide informed consent
* Clinically evaluated for need for initiation of new treatment (in patients not on current treatment), initiation of change in current treatment, or addition of new treatment (to any current treatment) in the setting of fibrotic hypersensitivity pneumonitis (HSP) or idiopathic pulmonary fibrosis (IPF), per standard of clinical care at UW Health.
* Willing and able to undergo PET/MRI.
* Participants requiring intravenous (IV) conscious sedation for imaging are not eligible; participants requiring mild, oral anxiolytics for the clinical MRI will be allowed to participate as long as the following criteria are met:

  * The subject has their own prescription for the medication
  * Informed consent is obtained prior to the self-administration of this medication
  * They come to the research visit with a driver

Exclusion Criteria:

* Participant is unable or unwilling to provide informed consent
* Participant is pregnant
* Participant with contraindication(s) to or inability to undergo PET/MRI
* Participants with contraindications to GBCA will be asked to undergo research imaging without the use of contrast. Contraindications may be severe kidney disease or previously documented GFR < 30 ml/min/1.73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in FAPI uptake | Baseline to 6 months
  FAPI uptake of fibrotic lesions as measured by Standardized Uptake Value (SUV). SUV quantifies the tracer uptake, helping to differentiate between normal and abnormal tissues and assess the extent of tumor activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Pirasteh, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No